CLINICAL TRIAL: NCT01752374
Title: Palonestron, Granisetron and Ramosetron for Prevention of Postoperative Nasea and Voming After Laparoscopic Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Won-Suk Lee, Prof, Gachon University Gil Medical Center
Other Study IDs: GIRBA2493
Record Dates: First submitted 2012-12-16; First posted 2012-12-19 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Female Patients Undergoing Laparoscopic Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Palonosetron group: Patient recieving Palonosetron/granisetron and ramosetron
- Granisetron group
- Ramosetron group

SUMMARY:
We compared the prophylactic anti-emetic efficacy of ramosetron, a newly developed 5-HT3 antagonist, granisetron and ondansetron in patients at high-risk for postoperative nausea and vomiting after laparoscpic abdominal surgery.

This study was conducted to determine the efficacy of three 5-HT3 receptor antagonists in the prevention of PONV for laparoscopic surgery in patients receiving PCA IV.

DETAILED DESCRIPTION:
Occurrences of nausea and vomiting, the severity of nausea (VAS), rescue antiemetic drug use, and amount of PCEA infusion and rescue pethidine were monitored after the end of surgery during four time periods: 0-2 h; 2-6 h; 6-24 h; and 24-48 h. Nausea was defined as the subjectively unpleasant sensation associated with awareness of the urge to vomit; vomiting included retching (defined as the laboured spastic, rhythmic contraction of the respiratory muscles without the expulsion of the gastric contents) and vomiting (defined as the forceful expulsion of gastric contents from the mouth) [11]. A complete response was defined as no PONV and no need for rescue anti-emetic drug. If two or more episodes of PONV occurred during the study period, a rescue anti-emetic (metoclopramide 10 mg) was given IV. The primary outcome was the incidence of nausea during the study period.

ELIGIBILITY:
Inclusion Criteria:

* female gender, non-smoking and use of postoperative opioids undergoing laparocopic abdominal surgery

Exclusion criteria included laparoscopic abdominal surgey, allergy to one of the study drugs, opioid dependence, history of gastro-intestinal disease or Parkinson's disease, history of previous PONV and motion sickness, contra-indication for epidural block (previous back surgery, bleeding diathesis or neurological dysfunction), anti-emetic medication within 24 h before surgery, inability to use the PCEA device or comprehend the visual analogue scales (VAS) for pain and nausea assessment, or unwillingness to be enrolled in the study.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size was determined based on the ability to detect a difference in the primary outcome variable, the incidence of nausea. With 30 patients in each group there was 80% power at an a of 0.05 to detect a 30% difference in the number of patients with nausea up to 24 h after surgery.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
severity of nasea | immediated postop to 48hrs after surgery

SECONDARY OUTCOMES:
frequency of rescue drug needed | postop to 48hrs after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Won-Suk Lee, Incheon, Incehon, South Korea

REFERENCES:
- [Background] Yoo JY, Chae YJ, Cho HB, Park KH, Kim JS, Lee SY. Comparison of the incidence of postoperative nausea and vomiting between women undergoing open or robot-assisted thyroidectomy. Surg Endosc. 2013 Apr;27(4):1321-5. doi: 10.1007/s00464-012-2607-7. Epub 2012 Dec 13. PMID 23239293
- [Derived] Lee WS, Lee KB, Lim S, Chang YG. Comparison of palonosetron, granisetron, and ramosetron for the prevention of postoperative nausea and vomiting after laparoscopic gynecologic surgery: a prospective randomized trial. BMC Anesthesiol. 2015 Sep 3;15:121. doi: 10.1186/s12871-015-0102-0. PMID 26335706